CLINICAL TRIAL: NCT02925416
Title: A Double-Blind, Randomized Study to Evaluate the Safety of Either a Single 1200-mg Intravenous (IV) Dose of Orbactiv™ (Oritavancin) and Placebo or Two IV Doses of Orbactiv™ in Subjects Being Treated for Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Brief Title: Safety of Either a Single or Two Intravenous Doses of Orbactiv in Participants With Acute Bacterial Skin and Skin Structure Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MDCO-ORI-16-02
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Skin Diseases, Bacterial
MeSH Terms: conditions — Skin Diseases, Bacterial | interventions — oritavancin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oritavancin/Oritavancin (Experimental): On Day 1, participants were administered a single 1200-mg IV dose of oritavancin in 1000 milliliters (mL) diluted in 5% dextrose in water (D5W). On Day 7, an additional 1200-mg IV dose of oritavancin in 1000 mL of D5W was administered.
  Interventions: Drug: Oritavancin
- Oritavancin/Placebo (Other): On Day 1, participants were administered a single 1200-mg IV dose of oritavancin in 1000 mL of D5W. On Day 7, a placebo was administered IV in 1000 mL of D5W.
  Interventions: Drug: Oritavancin; Drug: Placebo (D5W)

INTERVENTIONS:
Drug: Oritavancin — Administered intravenously
  Other Names: Orbactiv
Drug: Placebo (D5W) — Administered intravenously
  Arms: Oritavancin/Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of two 1200 milligram (mg) intravenous (IV) infusions of oritavancin when administered one week apart.

DETAILED DESCRIPTION:
Clinical studies in adult participants with acute bacterial skin and skin structure infection (ABSSSI) have demonstrated that a single 1200-mg IV dose of oritavancin was clinically non-inferior, well tolerated, and had a similar safety profile to 7 to 10 days of IV vancomycin treatment. The 1200-mg dose of oritavancin is the United States approved therapeutic dose.

Participants with ABSSSI were enrolled in this study to obtain safety information of two 1200-mg IV infusions of oritavancin when administered one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ABSSSI (wound infections, cellulitis/erysipelas, or cutaneous abscess) suspected or confirmed to be caused by a Gram-positive pathogen requiring IV therapy
* Able to give informed consent and willing to comply with all required study procedures

Exclusion Criteria:

* Infections associated with, or in close proximity to, a prosthetic device
* Severe sepsis or refractory shock
* Known or suspected bacteremia at time of screening
* ABSSSI due to or associated with any of the following:

  * Infections suspected or documented to be caused by Gram-negative pathogens (i.e., human or animal bites, injuries contaminated with fresh or salt water, external malignant otitis)
  * Wound infections (surgical or traumatic) and abscesses with only Gram-negative pathogens
  * Diabetic foot infections (infection extending distal to the malleoli in a participant with diabetes mellitus and peripheral neuropathy and/or vascular insufficiency or any ulceration of their foot)
  * Concomitant infection at another site not including a secondary ABSSSI lesion (e.g., septic arthritis, endocarditis, osteomyelitis)
  * Infected burns
  * A primary infection secondary to a pre-existing skin disease with associated inflammatory changes such as atopic dermatitis, eczema, or hidradenitis suppurativa
  * Decubitus or chronic skin ulcer, or ischemic ulcer due to peripheral vascular disease (arterial or venous)
  * Any evolving necrotizing process (i.e., necrotizing fasciitis), gangrene, or infection suspected or proven to be caused by Clostridium species (e.g., crepitance on examination of the ABSSSI site and/or surrounding tissue(s) or radiographic evidence of subcutaneous gas in proximity to the infection)
  * Infections known to be caused by a Gram-positive organism with a vancomycin minimum inhibitory concentration (MIC) >2 μg/mL or clinically failing prior therapy with glycopeptides
  * Catheter site infections
* Currently receiving chronic systemic immunosuppressive therapy such as chemotherapy or prednisone (prednisone at non-immunosuppressive doses of ≤15 mg/day is permitted)
* Participants who are likely to need treatment with IV unfractionated heparin sodium within 48 hours after oritavancin administration
* Last known cluster of differentiation 4 (CD4) count <200 cells/mm^3 in participants with known human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS)
* Neutropenia with absolute neutrophil count (ANC) <500 cells/mm^3
* Significant or life-threatening condition (e.g., endocarditis) that would confound or interfere with the assessment of safety
* Women who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least 2 acceptable methods of birth control: (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier method(s) or male partner sterilization). Women ≥2 years postmenopausal or surgically sterile are exempt from this exclusion
* History of immune-related hypersensitivity reaction to glycopeptides (such as vancomycin, televancin, daptomycin, or dalbavancin) or any of their excipients. Note: participants who have had histamine-like infusion reactions to a glycopeptide are not excluded
* Participants unwilling to forego blood and/or blood product donation for at least 1 month from initiation of oritavancin dose
* Treatment with investigational medicinal product within 30 days or 5 half-lives, whichever is longer, before enrollment and for the duration of the study
* Investigational device present, or removed within 30 days before enrollment, or presence of device-related infection
* Participants who the investigator considers unlikely to adhere to the protocol, comply with oritavancin administration, or complete the clinical study (e.g., unlikely to survive 90 days from initiation of oritavancin dosing)
* Prior exposure to oritavancin alone or in combination with another product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- South Jersey Infectious Disease, Somers Point, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oritavancin/Oritavancin: Participants received an intravenous (IV) infusion of 1200 milligrams (mg) of oritavancin on Day 1 and Day 7
- Oritavancin/Placebo: Participants received an IV infusion of 1200 mg of oritavancin on Day 1 and placebo on Day 7
Period: Overall Study
Arm/Group | Oritavancin/Oritavancin | Oritavancin/Placebo
Started | 17 | 5
Received at Least 1 Dose of Study Drug | 17 | 5
Completed | 15 | 5
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included participants who were screened and randomized
Groups:
- Oritavancin/Oritavancin: Participants received an IV infusion of 1200 mg of oritavancin on Day 1 and Day 7
- Total: Total of all reporting groups
Arm/Group | Oritavancin/Oritavancin | Oritavancin/Placebo | Total
Number analyzed (Participants) | 17 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 2 | 14
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 5 | 20
  Black or African American | 2 | 0 | 2
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment, including abnormal vital signs or laboratory assessments. Treatment emergent adverse events (TEAE) were AEs which occurred or whose severities worsened on or after the initiation of study drug. An SAE was defined as any untoward medical occurrence that at any dose resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 21 after first administration of oritavancin
Population: Safety population included all participants who were dosed with a dose of IV oritavancin
Measure: Count of Participants; unit: Participants
Arm/Group | Oritavancin/Oritavancin | Oritavancin/Placebo
Number analyzed (Participants) | 17 | 5
Participants
  At least 1 TEAE | 16 | 4
  At least 1 SAE | 0 | 0

2. Secondary Outcome: Number of Participants With a Clinical Response of Cure
Description: Participants were classified by investigator assessment as "success" for clinical response of cure if there was a complete or nearly complete resolution of baseline signs and symptoms of the primary infection such that no further treatment with antibiotics was needed.
Time Frame: Up to Day 8 after first administration of oritavancin
Population: Safety population included all participants who were dosed with a dose of IV oritavancin
Measure: Count of Participants; unit: Participants
Arm/Group | Oritavancin/Oritavancin | Oritavancin/Placebo
Number analyzed (Participants) | 17 | 5
Participants | 15 | 5

ADVERSE EVENTS:
Time Frame: Up to Day 21 after first administration of oritavancin
Description: Safety population included all participants who were dosed with a dose of IV oritavancin
Arm/Group | Oritavancin/Oritavancin | Oritavancin/Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/5
Other Adverse Events (participants affected / at risk) | 14/17 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oritavancin/Oritavancin (N=17) | Oritavancin/Placebo (N=5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Pyrexia (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Infusion Site Extravasation (General disorders) | 1 | 0
Skin Infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Rash Pustular (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Blood Pressure Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Blood Immunoglobulin E Increased (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT02925416/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02925416/SAP_001.pdf